CLINICAL TRIAL: NCT03490565
Title: PREoperativ Study of Exercise Training-RCT: A Phase 3 Randomized Controlled Trial of Preoperative Exercise Training vs Usual Care During Neoadjuvant Treatment in Patients With Gastroesophageal Cancer
Brief Title: PREoperativ Study of Exercise Training
Acronym: PRESET-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jesper Frank Christensen, PhD (Other)
Collaborators: Lundbeck Foundation (Other); Beckett Foundation (Other); Region Capital Denmark (Other)
Responsible Party: Sponsor-Investigator, Jesper Frank Christensen, PhD, Postdoc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRESET-RCT
Record Dates: First submitted 2018-03-23; First posted 2018-04-06 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: GastroEsophageal Cancer
Keywords: exercise training; treatment tolerability; treatment complications
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EX group (Active Comparator): Exercise training
  Interventions: Behavioral: Exercise training
- CON-group (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Exercise training — Structured, supervised, high-intensity combined aerobic and resistance exercise. Based on patients' individual capacity (Wattmax and 1RM), a personalized exercise program will be prescribed. Following a 5 minutes warm up, the patients will perform 21 min of aerobic interval training on a stationary bicycle consisting of three 4 minute high intensity intervals (85-95% HRmax) with 3 minutes of active pause between each interval. The resistance training comprises 4 functional exercises by performed using bodyweight, elastic resistance bands or kettlebells followed by resistance exercises in machines for the major muscle groups: chest press, leg press, seated rows, and leg extension with 1 warm-up set followed by 3-4 sets of 8 to 12 repetitions.
  Arms: EX group

SUMMARY:
Background Patients undergoing resection for gastro-esophageal (GE)-cancer are subjected to high burden of disease and treatment-specific morbidities with potential detrimental impact on survival and quality of life. Exercise training is a promising strategy to improve physical functional before and after tumor resection, but it is not established if this translates into lower risk of peri- and post-operative complications, improved treatment tolerance.

Objectives:

* To explore the effect a preoperative exercise-training intervention on the risk of treatment failure, defined as the risk of not reaching surgery, in patients diagnosed with operable GE cancer.
* To explore the effect of preoperative exercise training on median time to tumor progression (disease free survival), and overall survival
* To explore the effect of preoperative exercise training on the risk of treatment complications
* To explore the effect of preoperative exercise training on health related quality of life, anxiety and depression,cardiopulmonary fitness, muscle strength, and body composition

Subjects and Methods In total, 310 GE-cancer patients will be included in the study and randomly allocated to pre-operative exercise training (n=155) or usual care control (n=155). All participants will undergo 2 study visits; assessed for cardiopulmonary fitness; muscle strength, body composition; blood sample (50 ml); quality of life by questionnaires; physical function; and blood volume profile.

Quality of life will be assessed by questionnaires by self-report three times (at 12, 24, and 36 months after diagnosis), and we will collect data from medical records regarding mortality and disease recurrence up to 36 months after diagnosis.

Treatment arms:

The intervention-group will be prescribed 2-3 weekly supervised exercise training for a total of 12 weeks before surgery during neo-adjuvant chemotherapy. The control group will follow current usual care guidelines. After surgery during adjuvant chemotherapy, both groups will be referred to municipality-based rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically verified, resectable adenocarcinoma of the esophagus, stomach or gastro-esophageal junction

Exclusion Criteria:

* Deemed inoperable at the point of diagnoses
* Pregnancy
* Any other known malignancy requiring active treatment
* Not eligible for preoperative chemo- or chemoradiotherapy
* Performance status > 1
* Physical disabilities precluding physical testing and/or exercise
* Inability to read and understand Danish

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of treatment failure | From date of randomization, until the date of treatment failure is clinically determined before scheduled surgery assessed for up to 20 weeks
  The frequency of patients scheduled to receive neo-adjuvant treatment and tumor resection with curative intend, but fail to reach surgery due to death, disease progression or physical deterioration

SECONDARY OUTCOMES:
Time to disease progression | Baseline to 3 year follow-up
  Time from point of diagnosis to clinical disease relapse
3 year disease free survival | Baseline to 3 year follow-up
  Frequency of patients alive without clinical disease relapse 3 years after diagnosis
3 year overall survival | Baseline to 3 year follow-up
  Frequency of patients alive 3 years after diagnosis
Health Related Quality of Life | Baseline, scheduled surgery, 1-year follow-up, 2-year follow-up, 3-year follow-up
  Changes from baseline in the Functional Assessment of Cancer Therapy (FACT) questionaire
Anxiety and Depression | Baseline, scheduled surgery, 1-year follow-up, 2-year follow-up, 3-year follow-up
  Changes from baseline in the HADs questionaire
Pre-operative risk of hospitalization | From date of randomization, until the date of hospitilization before scheduled surgery assessed for up to 20 weeks
  Frequency of non-scheduled hospitalization during neoadjuvant treatment
Total length of hospital stays | From date of randomization up to 30 days after surgery
  Total number of days hospitalized
Tumor regression grade | From date of randomization (baseline tumor biopsy) to tumor resection (surgery), up to 20 weeks
  Pathology assessment of tumor response to neoadjuvant treatment
Risk of neoadjuvant treatment dose-reduction | From date of randomization to the date of surgery, up to 20 weeks
  Incidence of dose-reduction
Risk of neoadjuvant treatment complications | From date of randomization to the date of surgery, up to 20 weeks
  Incidence of registered toxicities (graded 1-4)
Risk of post-operative complications | From surgery to 30 days post surgery
  Incidence of registered post-operative complications (Clavien-Dindo grade 2-4)
Cardiopulmonary fitness | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in VO2peak
Maximum muscle strength | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in 1 repetition maximum strength leg-press
Lean Body Mass | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in whole-body lean mass assessed by
  dual energy x-ray absorptiometry (DXA) scan
Fat percentage | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in whole-body fat percentage assessed by DXA scan
Appendicular lean mass | Baseline to scheduled surgery
  Changes in appendicular lean mass assessed by DXA scan
Leg-extensor power | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in maximum leg power assessed by Nottingham Power Rig
Blood Volume | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in blood volume assessed by CO2 rebreathing
TNFa | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in plasma TNFa concentration
Interleukin (IL)-6 | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in plasma IL-6 concentration
CRP | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in plasma CRP concentration
HbA1c | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in plasma HbA1c concentration
IL-10 | From visit 1 (date of randomization, before neoajuvant treatment) until to visit 2 (the week before surgery, after neoadjuvant treatment) up to 20 weeks
  Changes in plasma IL-10 concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jesper F Christensen, PhD, Principal Investigator — Rigshospitalet, Denmark; Lars B Svendsen, DMSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No